CLINICAL TRIAL: NCT06440356
Title: Effect of Non-invasive Photobiomodulation Therapies in Patients With Trigeminal Neuralgia: A Randomised, Placebo-controlled Trial
Brief Title: Effect of Non-invasive Photobiomodulation Therapies in Patients With Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, İREM KARAGOZOGLU, Assist. Prof., University of Gaziantep
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UGaziantep1986
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment protocol (Experimental): In the first group, a NGD laser with dual wavelength, infrared and LED features, operating at a depth of 50 mm, which can be applied regionally, was used.
  In the second group, a neodymium-doped yttrium aluminium garnet laser was used. After the laser unit has been switched on, the LLLT preset has been selected.
  Patients in the third group received emission-free laser treatment. In the same procedure with the Nd:YAG laser, a placebo treatment was performed with the device on, laser beams visible but not active.
  Interventions: Other: laser therapy

INTERVENTIONS:
Other: laser therapy — low level laser therapy applied

SUMMARY:
The aim of this study was to compare the effectiveness of two different photobiomodulation (PBM) therapies as an alternative to medical treatment to reduce pain and improve quality of life in patients with trigeminal neuralgia (TN).

DETAILED DESCRIPTION:
The aim of this study was to compare the effectiveness of two different photobiomodulation (PBM) therapies as an alternative to medical treatment to reduce pain and improve quality of life in patients with trigeminal neuralgia (TN). A total of 45 patients with mean age of 46.09 years (26 female, 19 male) were randomly divided into three groups. The first group received PBM therapy with a new generation diode laser (NGD laser). In the second group, low-level Nd:YAG laser was applied along the affected nerve line and the placebo group received the same protocol with Nd:YAG laser without the device switched on. The scores were recorded before and after the treatment using the Brief Pain Inventory-facial (BPI-facial) scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic trigeminal neuralgia as defined by the International Headache Society (2).
* Patients diagnosed with idiopathic trigeminal neuralgia and receiving medical treatment (carbamazepine, etc.)
* Patients with unilateral, severe, sudden onset of facial pain along the branches of the trigeminal nerve.
* Patients who have not previously received any interventional treatment for TN.
* Patients recently diagnosed and started on a first dose of carbamazepine and its derivatives

Exclusion Criteria:

* • Patients diagnosed with type 2 (atypical, symptomatic) trigeminal neuralgia as defined by the International Headache Society (2).

  * Patients with etiologies such as tumour, multiple sclerosis or neurovascular compression on radiography.
  * Pregnant women
  * Patients with systemic diseases such as diabetes, cardiovascular disease, hypertension, etc.
  * Patients who have been previously diagnosed and treated with any type of TN therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain intensity on the 10 point Brief Pain Inventory-facial scale at week 4. | baseline and week 4
  Brief Pain Inventory-facial scale is a validated, self-reported scale assessing the average pain intensity over the past 24 hour period. The scores range from 0: no pain, 10: the worst pain you can imagine change= week 4 score-baseline score
Change from baseline in interference in general activities on the 10 point Brief Pain Inventory-facial scale at week 4. | baseline and week 4
  Brief Pain Inventory-facial scale is a validated, self-reported scale assessing the interference in general activities over the past 24 hour period. The scores range from 0: no inhibition, 10: complete inhibition change= week 4 score-baseline score

SECONDARY OUTCOMES:
Change from baseline in interference in face specific activities on the 10 point Brief Pain Inventory-facial scale at week 4. | baseline and week 4
  Brief Pain Inventory-facial scale is a validated, self-reported scale assessing the interference in face specific activities over the past 24 hour period. The scores range from 0: no inhibition, 10: complete inhibition change= week 4 score-baseline score

CONTACTS AND LOCATIONS:
Locations (1):
- İrem Karagözoğlu, Şehitkamil, Gazi̇antep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No